CLINICAL TRIAL: NCT05920200
Title: Factors Affecting the Results of Treatment of Patients With Hernias of Various Localization: Evaluation of Treatment Results Using an Automated Hernia Register
Brief Title: Factors Influencing the Results of Treatment in Patients With Hernias of Various Localizations
Status: Recruiting | Type: Observational
Sponsor: Immanuel Kant Baltic Federal University (Other)
Responsible Party: Sponsor
Other Study IDs: HR202339
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Inguinal Hernia; Femoral Hernia; Umbilical Hernia; Ventral Hernia; Chronic Pain; Acute Post Operative Pain; Recrrence Rate
Keywords: hernia; register; inguinal hernia; femoral hernia; umbilical hernia; ventral hernia; CPIP; postoperative complications; chronic post-operative pain; recurrence rate
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Hernia, Umbilical; Hernia, Ventral; Chronic Pain; Pain, Postoperative; Hernia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with groin and femoral hernia/IG
  Interventions: Procedure: open non-mesh hernia repair; Procedure: open mesh hernia repair; Procedure: MIS hernia repair
- Patients with umbilical hernia/IG
  Interventions: Procedure: open non-mesh hernia repair; Procedure: open mesh hernia repair; Procedure: MIS hernia repair
- Patients with ventral and incisional hernia/InG
  Interventions: Procedure: open non-mesh hernia repair; Procedure: open mesh hernia repair; Procedure: MIS hernia repair

INTERVENTIONS:
Procedure: open non-mesh hernia repair — A groin and femoral hernia non-mesh repair. An umbilical hernia non-mesh repair. A ventral and incisional hernia non-mesh repair.
Procedure: open mesh hernia repair — A groin and femoral hernia repair, reinforced by synthetic mesh. The mesh is affixed with sutures for Lichtenstein. Self-fixating mesh is also possible.
  An umbilical, ventral, incisional hernia repair, reinforced by synthetic mesh. The mesh is affixed with sutures.
Procedure: MIS hernia repair — A groin and femoral minimal invasive hernia repair (TAPP, eTEP). The mesh is affixed with tack/no-fixation. Self-fixation mesh is also possible.
  An umbilical, ventral, incisional minimal invasive hernia repair (eTEP, IPOM,). The mesh is affixed with tack and no-fixation .

SUMMARY:
The study attempts to quantify the relative risks for acute postoperative pain, complications rate, chronic postoperative pain (CPIP) and recurrence rate after different methods of repair of groin, umbilical and incisional hernia depending on surgical technique, mesh type and fixation suture material.

For this purpose the investigators will analyze data from the Kalinigrad Hernia Registry (KHR).

ELIGIBILITY:
Inclusion Criteria:

* All mesh and non-mesh repairs that have been registered in the KHR from January 9, 2020, until December 31, 2023.

Exclusion Criteria:

* Patients not having a 11-digit state-assigned Personal insurance policy number.
* Parastomal hernia;
* infected hernias;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An unselected, consecutive regionwide cohort during 3 years, with a 3-year follow-up
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic postoperative pain rate and severity | 1 year
  The painDETECT questionnaire will be used to identify chronic postoperative pain.
  Final painDETECT Score: 20, indicating that a neuropathic pain component is likely (>90%).
Recurrence rate | 3 year
  the overall frequency of recurrent hernias

SECONDARY OUTCOMES:
Treatment satisfaction rate | 3 year
  To assess the quality of life will be used Eura HS Quality of Life Scale-EuraHS QoL.
  EuraHS Qol - total (min - 0, max - 90) EuraHS Qol - pain (min - 0, max - 30) EuraHS Qol - restriction of activities (min - 0, max - 40) EuraHS Qol - cosmetic discomfort (min -0, max - 20)
  Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Baltic Federal University, Kaliningrad, Kaliningrad Oblast, Russia

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be available for other researcher.